CLINICAL TRIAL: NCT02404844
Title: Molecularly Stratified Parallel Cohort, Single Arm Phase II Trial of the Phosphoinositide 3-kinase (PI3K) Inhibitor Buparlisib (BKM120) in Combination With Tamoxifen in Patients With Hormone Receptor-positive, HER2-negative Inoperable (Locally Advanced or Metastatic) Breast Cancer With Prior Exposure to Antihormonal Therapy
Brief Title: Trial of BKM120/Tamoxifen-combination in Patients With HR-pos, HER2-neg Breast Cancer
Acronym: PIKTAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Collaborators: iOMEDICO AG (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Anja Welt, Principal Investigator, University Hospital, Essen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iOM-02282; 2014-000599-24 (EudraCT Number); CBKM120ZDE02T (Other Grant/Funding Number: Novartis Pharma GmbH); AIO-MAM-0114/ass (Other Grant/Funding Number: AIO)
Record Dates: First submitted 2015-02-20; First posted 2015-04-01 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — NVP-BKM120; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BKM120 + Tamoxifen (Experimental): BKM120 (Buparlisib): 100 mg/day, orally, on a continuous dosing schedule without interruption starting on day 1 in 28 day cycle
  Tamoxifen: 20 mg/day, orally, on a continuous dosing schedule without interruption starting on day 1 in 28 day cycle
  Interventions: Drug: BKM120; Drug: Tamoxifen

INTERVENTIONS:
Drug: BKM120 — daily oral
  Other Names: Buparlisib
Drug: Tamoxifen — daily oral

SUMMARY:
This is a clinical trial with a molecularly stratified parallel cohort, single arm design to explore the efficacy and safety of BKM120 in combination with tamoxifen in patients with ER/PR-positive, HER2-negative breast cancer with prior exposure to antihormonal therapy, and different biomarker profiles, two of them potentially indicative of constitutive PI3K pathway activation.

DETAILED DESCRIPTION:
This is a clinical trial with a molecularly stratified parallel cohort, single arm design to explore the efficacy and safety of BKM120 in combination with tamoxifen in patients with ER/PR-positive, HER2-negative breast cancer with prior exposure to antihormonal therapy, and different biomarker profiles, two of them potentially indicative of constitutive PI3K pathway activation:

* PIK3CA mutation/preserved PTEN expression
* PIK3CA wildtype or mutation/ loss of PTEN expression
* PIK3CA wildtype/preserved PTEN expression. This trial will explore, if the combination of BKM120 and tamoxifen can overcome resistance to antihormonal therapies. BKM120 is selective for class I PI3K enzymes with no mTOR inhibitory activity that has entered Phase II and III clinical trials. The tumor suppressor PTEN is the most important negative regulator of the PI3K signaling pathway. Therefore, in addition the trial will prospectively evaluate PIK3CA mutations and/or loss of PTEN expression as predictive biomarkers for clinical benefit from combined treatment with BKM120 and tamoxifen.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically and/or cytologically confirmed diagnosis of breast cancer
* Patient has radiologic or objective evidence of inoperable locally advanced, or metastatic breast cancer
* Patient has a known hormone receptor status HR-positive (ER and/or PR positive) and HER2-negative status
* Patient has a representative archival formalin-fixed tumor biopsy (metastasis or primary tumor)
* Patient has prior exposure to antihormonal therapy
* Patient has received ≤ 2 prior antihormonal treatments in the metastatic setting
* Prior treatment with tamoxifen in the (neo-)adjuvant setting is allowed but has to be discontinued for at least 1 year.
* Patient may have received up to one prior chemotherapy in the metastatic setting
* Measurable or non-measurable lesions according to RECIST v1.1 criteria
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2

Exclusion Criteria:

* Patient has received previous treatment with a PI3K- or AKT-inhibitor or mTOR-inhibitors
* Prior treatment with Tamoxifen in the metastatic setting. Treatment with tamoxifen in the (neo-)adjuvant setting is allowed, but has to be discontinued for at least 1 year
* Patient has symptomatic CNS metastases
* Patient has a medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others), or patients with active severe personality disorders (defined according to DSM-IV).
* Patient has a known history of HIV infection (testing not mandatory) infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12; Primary Completion 2017-09-19 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS)-rate in the full population, after 6 months | 6 months
  PFS is defined as time from date of start of treatment to the date of the event, defined as the first documented disease progression or death due to any cause per local investigator assessment

SECONDARY OUTCOMES:
Progression free survival (PFS)- rate in the subpopulations after 6 months of combination therapy | 6 months
  PFS is defined as time from date of start of treatment to the date of the event, defined as the first documented disease progression or death due to any cause per local investigator assessment
Progression-free survival (PFS) | 6 months
  PFS in subpopulations and full population. PFS is defined as time from date of start of treatment to the date of the event, defined as the first documented disease progression or death due to any cause per local investigator assessment
1 year overall survival (OS) rate | 1 year
  OS is defined as time from date of start of treatment to the date of death from any cause.
2 years overall survival (OS) rate | 2 years
  OS is defined as time from date of start of treatment to the date of death from any cause.
Overall response rate (ORR) | 6 months
  ORR is defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) (RECIST v1.1).
Disease control rate (DCR) | 6 months
  DCR is defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) or stable disease (SD) lasting more than 12 weeks (RECIST v1.1).
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From date of informed consent to +30 days from last application of study medication
  Type, frequency and severity of adverse events per CTCAE v4.03
Incidence and severity of depressive episodes during the course of treatment | From date of informed consent to +30 days from last application of study medication
  Change in depressive episodes assessed by PHQ-9 questionnaire
Incidence and severity of depressive episodes during the course of treatment | From date of informed consent to +30 days from last application of study medication
  Change in depressive episodes assessed by GAD-7 questionnaire

OTHER OUTCOMES:
Identification of genomic signatures associated with clinical outcome in response to PI3K pathway-directed therapy with tamoxifen and buparlisib in ER/PR-positive breast cancer. | 2 years
  Finding of genomic signatures associated with clinical outcome in response to PI3K pathway-directed therapy with tamoxifen and buparlisib in ER/PR-positive breast cancer.
Validation of a proprietary technology for highly sensitive and specific mutation detection of circulating free tumor DNA | 2 years
  Finding of specific mutation detection of circulating free tumor DNA

CONTACTS AND LOCATIONS:
Overall Officials: Anja Welt, MD, Principal Investigator — University Hospital, Essen
Locations (1):
- iOMEDICO AG, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Bendell JC, Rodon J, Burris HA, de Jonge M, Verweij J, Birle D, Demanse D, De Buck SS, Ru QC, Peters M, Goldbrunner M, Baselga J. Phase I, dose-escalation study of BKM120, an oral pan-Class I PI3K inhibitor, in patients with advanced solid tumors. J Clin Oncol. 2012 Jan 20;30(3):282-90. doi: 10.1200/JCO.2011.36.1360. Epub 2011 Dec 12. PMID 22162589
- [Background] Rodon J, Brana I, Siu LL, De Jonge MJ, Homji N, Mills D, Di Tomaso E, Sarr C, Trandafir L, Massacesi C, Eskens F, Bendell JC. Phase I dose-escalation and -expansion study of buparlisib (BKM120), an oral pan-Class I PI3K inhibitor, in patients with advanced solid tumors. Invest New Drugs. 2014 Aug;32(4):670-81. doi: 10.1007/s10637-014-0082-9. Epub 2014 Mar 21. PMID 24652201